CLINICAL TRIAL: NCT00583908
Title: Clinical and Theoretical Evaluation of Factors Affecting Soft Toric Lens Performance: Part 3
Brief Title: Evaluation of Orientation and Visual Acuity of Four Toric Soft Contact Lenses When Head is Tilted at 90 Degrees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Collaborators: Visioncare Research Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-0710 pt 3; ETOR-507(under GNR-011)
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Results first posted 2009-09-28 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Astigmatism
Keywords: astigmatism; orientation; visual acuity; contact lenses
MeSH Terms: conditions — Astigmatism; Orientation, Spatial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (12):
- Group 1: lotrafilcon B/senofilcon A/balafilcon A/omafilcon A (Active Comparator): One intervention was worn during each study period, which consisted of lens insertion, followed by a 15 minute settling period prior to measurement. All four periods were conducted in one day. Period 1: lotrafilcon B /period 2: senofilcon A / period 3: balafilcon A / period 4: omafilcon A
  Interventions: Device: senofilcon A; Device: balafilcon A toric; Device: lotrafilcon B toric; Device: omafilcon A
- Group 2 lotrafilcon B/omafilcon A/senofilcon A/balafilcon A (Active Comparator): One intervention was worn during each study period, which consisted of lens insertion, followed by a 15 minute settling period prior to measurement. All four periods were conducted in one day. period 1: lotrafilcon B / period 2: omafilcon A / period 3: senofilcon A / period 4: balafilcon A
  Interventions: Device: senofilcon A; Device: balafilcon A toric; Device: lotrafilcon B toric; Device: omafilcon A
- Group 3 lotrafilcon B/balafilcon A/senofilcon A/omafilcon A (Active Comparator): One intervention was worn during each study period, which consisted of lens insertion, followed by a 15 minute settling period prior to measurement. All four periods were conducted in one day. period 1: lotrafilcon B / period 2: balafilcon A / period 3: senofilcon A / period 4: omafilcon A
  Interventions: Device: senofilcon A; Device: balafilcon A toric; Device: lotrafilcon B toric; Device: omafilcon A
- Group 4 senofilcon A/lotrafilcon B/omafilcon A/balafilcon A (Active Comparator): One intervention was worn during each study period, which consisted of lens insertion, followed by a 15 minute settling period prior to measurement. All four periods were conducted in one day. period 1: senofilcon A / period 2: lotrafilcon B / period 3: omafilcon A / period 4: balafilcon A
  Interventions: Device: senofilcon A; Device: balafilcon A toric; Device: lotrafilcon B toric; Device: omafilcon A
- Group 5 senofilcon A/omafilcon A/balafilcon A/lotrafilcon B (Active Comparator): One intervention was worn during each study period, which consisted of lens insertion, followed by a 15 minute settling period prior to measurement. All four periods were conducted in one day. period 1: senofilcon A / period 2: omafilcon A / period 3: balafilcon A / period 4: lotrafilcon B
  Interventions: Device: senofilcon A; Device: balafilcon A toric; Device: lotrafilcon B toric; Device: omafilcon A
- Group 6 senofilcon A/balafilcon A/lotrafilcon B/omafilcon A (Active Comparator): One intervention was worn during each study period, which consisted of lens insertion, followed by a 15 minute settling period prior to measurement. All four periods were conducted in one day. period 1: senofilcon A / period 2: balafilcon A / period 3: lotrafilcon B / period 4: omafilcon A
  Interventions: Device: senofilcon A; Device: balafilcon A toric; Device: lotrafilcon B toric; Device: omafilcon A
- Group 7 omafilcon B/lotrafilcon B/senofilcon A/balafilcon A (Active Comparator): One intervention was worn during each study period, which consisted of lens insertion, followed by a 15 minute settling period prior to measurement. All four periods were conducted in one day. period 1: omafilcon A / period 2: lotrafilcon B / period 3: senofilcon A / period 4: balafilcon A
  Interventions: Device: senofilcon A; Device: balafilcon A toric; Device: lotrafilcon B toric; Device: omafilcon A
- Group 8 balafilcon A/lotrafilcon B/senofilcon A/omafilcon A (Active Comparator): One intervention was worn during each study period, which consisted of lens insertion, followed by a 15 minute settling period prior to measurement. All four periods were conducted in one day. period 1: balafilcon A / period 2: lotrafilcon B / period 3: senofilcon A / period 4: omafilcon A
  Interventions: Device: senofilcon A; Device: balafilcon A toric; Device: lotrafilcon B toric; Device: omafilcon A
- Group 9 balafilcon A/lotrafilcon B/omafilcon A/senofilcon A (Active Comparator): One intervention was worn during each study period, which consisted of lens insertion, followed by a 15 minute settling period prior to measurement. All four periods were conducted in one day. period 1: balafilcon A / period 2: lotrafilcon B / period 3: omafilcon A / period 4: senofilcon A
  Interventions: Device: senofilcon A; Device: balafilcon A toric; Device: lotrafilcon B toric; Device: omafilcon A
- Group 10 balafilcon A/senofilcon A/lotrafilcon B/omafilcon A (Active Comparator): One intervention was worn during each study period, which consisted of lens insertion, followed by a 15 minute settling period prior to measurement. All four periods were conducted in one day. period 1: balafilcon A / period 2: senofilcon A / period 3: lotrafilcon B / period 4: omafilcon A
  Interventions: Device: senofilcon A; Device: balafilcon A toric; Device: lotrafilcon B toric; Device: omafilcon A
- Group 11 balafilcon A/senofilcon A/omafilcon A//lotrafilcon B (Active Comparator): One intervention was worn during each study period, which consisted of lens insertion, followed by a 15 minute settling period prior to measurement. All four periods were conducted in one day. period 1: balafilcon A / period 2: senofilcon A / period 3: omafilcon A / period 4: lotrafilcon B
  Interventions: Device: senofilcon A; Device: balafilcon A toric; Device: lotrafilcon B toric; Device: omafilcon A
- Group 12 balafilcon A/omafilcon A/lotrafilcon B/senofilcon A (Active Comparator): One intervention was worn during each study period, which consisted of lens insertion, followed by a 15 minute settling period prior to measurement. All four periods were conducted in one day. period 1: balafilcon A / period 2: omafilcon A / period 3: lotrafilcon B / period 4: senofilcon A
  Interventions: Device: senofilcon A; Device: balafilcon A toric; Device: lotrafilcon B toric; Device: omafilcon A

INTERVENTIONS:
Device: senofilcon A — toric contact lens
Device: balafilcon A toric — toric contact lens
Device: lotrafilcon B toric — toric contact lens
Device: omafilcon A — toric contact lens

SUMMARY:
The purpose of this study is to determine the relative performance of a new toric soft contact lens against three toric contact lens currently available in market, specifically with orientation and visual acuity when head is tilted at 90 degrees.

DETAILED DESCRIPTION:
Non-dispensing single-masked (subject-masked), randomised, 1-visit controlled study, ~2 hour duration.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 and less than or equal to 50 years of age
2. be able and willing to adhere to the instructions set forth in the protocol.
3. have a distance spherical component between -1.00 D and -6.00D with cylinder in the range of 0.75 D to 1.75D
4. Sign the STATEMENT OF INFORMED CONSENT.
5. Have normal, healthy eyes

Exclusion Criteria:

1. The presence of ocular or systemic disease or need for medication which might interfere with contact lens wear.
2. Pre-existing ocular disease precluding contact lens fitting.
3. Insufficient lacrimal secretions
4. Aphakia, keratoconus or a highly irregular cornea
5. Previous eye surgery involving the anterior segment
6. Current pregnancy or lactation (to the best of the subject's knowledge).
7. Use of concurrent ocular medication
8. Active participation in another clinical study at any time during this study.-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2007-11; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Young, BSc, MPhil, Principal Investigator — Visioncare Research Ltd.
Locations (1):
- Visioncare Research Ltd., Farnham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Lotrafilcon B / Senofilcon A / Balafilcon A / Omafilcon A; Lotrafilcon B / Omafilcon A / Senofilcon A / Balafilcon A; Lotrafilcon B / Balafilcon A / Senofilcon A / Omafilcon A; Senofilcon A / Lotrafilcon B / Omafilcon A / Balafilcon A; Senofilcon A / Omafilcon A / Balafilcon A / Lotrafilcon B; Senofilcon A / Balafilcon A / Lotrafilcon B / Omafilcon A; Omafilcon A / Lotrafilcon B / Senofilcon A / Balafilcon A; Balafilcon A / Lotrafilcon B / Senofilcon A / Omafilcon A; Balafilcon A / Lotrafilcon B / Omafilcon A / Senofilcon A; Balafilcon A / Senofilcon A / Lotrafilcon B / Omafilcon A; Balafilcon A / Senofilcon A / Omafilcon A / Lotrafilcon A; Balafilcon A / Omafilcon A / Lotrafilcon B / Senofilcon A: All lenses were toric lenses. The order of lenses in the title relates to the period of administration.
Period: Period 1 - First Intervention
Arm/Group | Lotrafilcon B / Senofilcon A / Balafilcon A / Omafilcon A | Lotrafilcon B / Omafilcon A / Senofilcon A / Balafilcon A | Lotrafilcon B / Balafilcon A / Senofilcon A / Omafilcon A | Senofilcon A / Lotrafilcon B / Omafilcon A / Balafilcon A | Senofilcon A / Omafilcon A / Balafilcon A / Lotrafilcon B | Senofilcon A / Balafilcon A / Lotrafilcon B / Omafilcon A | Omafilcon A / Lotrafilcon B / Senofilcon A / Balafilcon A | Balafilcon A / Lotrafilcon B / Senofilcon A / Omafilcon A | Balafilcon A / Lotrafilcon B / Omafilcon A / Senofilcon A | Balafilcon A / Senofilcon A / Lotrafilcon B / Omafilcon A | Balafilcon A / Senofilcon A / Omafilcon A / Lotrafilcon A | Balafilcon A / Omafilcon A / Lotrafilcon B / Senofilcon A
Started | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 - Second Intervention
Arm/Group | Lotrafilcon B / Senofilcon A / Balafilcon A / Omafilcon A | Lotrafilcon B / Omafilcon A / Senofilcon A / Balafilcon A | Lotrafilcon B / Balafilcon A / Senofilcon A / Omafilcon A | Senofilcon A / Lotrafilcon B / Omafilcon A / Balafilcon A | Senofilcon A / Omafilcon A / Balafilcon A / Lotrafilcon B | Senofilcon A / Balafilcon A / Lotrafilcon B / Omafilcon A | Omafilcon A / Lotrafilcon B / Senofilcon A / Balafilcon A | Balafilcon A / Lotrafilcon B / Senofilcon A / Omafilcon A | Balafilcon A / Lotrafilcon B / Omafilcon A / Senofilcon A | Balafilcon A / Senofilcon A / Lotrafilcon B / Omafilcon A | Balafilcon A / Senofilcon A / Omafilcon A / Lotrafilcon A | Balafilcon A / Omafilcon A / Lotrafilcon B / Senofilcon A
Started | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 - Third Intervention
Arm/Group | Lotrafilcon B / Senofilcon A / Balafilcon A / Omafilcon A | Lotrafilcon B / Omafilcon A / Senofilcon A / Balafilcon A | Lotrafilcon B / Balafilcon A / Senofilcon A / Omafilcon A | Senofilcon A / Lotrafilcon B / Omafilcon A / Balafilcon A | Senofilcon A / Omafilcon A / Balafilcon A / Lotrafilcon B | Senofilcon A / Balafilcon A / Lotrafilcon B / Omafilcon A | Omafilcon A / Lotrafilcon B / Senofilcon A / Balafilcon A | Balafilcon A / Lotrafilcon B / Senofilcon A / Omafilcon A | Balafilcon A / Lotrafilcon B / Omafilcon A / Senofilcon A | Balafilcon A / Senofilcon A / Lotrafilcon B / Omafilcon A | Balafilcon A / Senofilcon A / Omafilcon A / Lotrafilcon A | Balafilcon A / Omafilcon A / Lotrafilcon B / Senofilcon A
Started | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 - Fourth Intervention
Arm/Group | Lotrafilcon B / Senofilcon A / Balafilcon A / Omafilcon A | Lotrafilcon B / Omafilcon A / Senofilcon A / Balafilcon A | Lotrafilcon B / Balafilcon A / Senofilcon A / Omafilcon A | Senofilcon A / Lotrafilcon B / Omafilcon A / Balafilcon A | Senofilcon A / Omafilcon A / Balafilcon A / Lotrafilcon B | Senofilcon A / Balafilcon A / Lotrafilcon B / Omafilcon A | Omafilcon A / Lotrafilcon B / Senofilcon A / Balafilcon A | Balafilcon A / Lotrafilcon B / Senofilcon A / Omafilcon A | Balafilcon A / Lotrafilcon B / Omafilcon A / Senofilcon A | Balafilcon A / Senofilcon A / Lotrafilcon B / Omafilcon A | Balafilcon A / Senofilcon A / Omafilcon A / Lotrafilcon A | Balafilcon A / Omafilcon A / Lotrafilcon B / Senofilcon A
Started | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study Population: Summary for overall study population
Arm/Group | Overall Study Population
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 5
Region of Enrollment [Number; unit: participants]
  United Kingdom | 14

OUTCOME MEASURES:

1. Primary Outcome: Lens Orientation During Head Tilt.
Description: Degree of lens rotation on the eye with the head tilted.
Time Frame: after fit of each of the four lens insertions
Population: Only participants who completed the study per protocol. Some participants had missing data for some lenses.
Measure: Mean (Standard Deviation); unit: Degree of rotation
Groups:
- Senofilcon A Toric: senofilcon A toric worn in either the first, second, third or fourth periods.
- Balafilcon A Toric: balafilcon A toric worn in either the first, second, third or fourth periods
- Lotrafilcon B Toric: lotrafilcon B toric worn in either the first, second, third, or fourth periods.
- Omafilcon A Toric: omafilcon A toric worn in either the first, second, third, or fourth periods.
Arm/Group | Senofilcon A Toric | Balafilcon A Toric | Lotrafilcon B Toric | Omafilcon A Toric
Number analyzed (Participants) | 13 | 13 | 13 | 11
Degree of rotation | 12.2 (10.7) | 39.7 (18.5) | 27.6 (22.7) | 39.3 (15.9)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Alternative Hypothesis was senofilcon A toric was superior to balafilcon A toric by having less degrees of rotation; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — Paired t-test; Mean Difference (Final Values) = -27.5, Standard Deviation 17.1 — mean difference was senofilcon A minus balafilcon A
Statistical Analysis 2: Comparison: Senofilcon A Toric vs Lotrafilcon B Toric; Hypothesis was senofilcon A toric was superior to lotrafilcon B toric by having less degree of rotation; Test type: Superiority or Other; p = 0.0002, t-test, 1 sided — paired t-test; Mean Difference (Final Values) = -15.4, Standard Deviation 17.8 — mean difference is senofilcon A minus lotrafilcon B
Statistical Analysis 3: Comparison: Senofilcon A Toric vs Omafilcon A Toric; Hypothesis was senofilcon A toric was superior to omafilcon A toric by having less degree of rotation; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided — paired t-test; Mean Difference (Final Values) = -27.0, Standard Deviation 12.4 — Mean difference is senofilcon A minus omafilcon A

2. Primary Outcome: Visual Acuity During Head Tilt
Description: logarithm of the minimum angle of resolution (logMar) ideal is 0.0 and represents 20/20 Snellen acuity.
  logMar values > 0.00 indicate vision poorer than the ideal and values <0.00 indicate vision greater than the ideal.
Time Frame: after each of the four lens insertions
Population: Only participants who completed the study per protocol. Some participants had missing data for some of the lenses.
Measure: Mean (Standard Deviation); unit: logMAR units
Arm/Group | Senofilcon A Toric | Balafilcon A Toric | Lotrafilcon B Toric | Omafilcon A Toric
Number analyzed (Participants) | 13 | 13 | 13 | 11
logMAR units | 0.02 (0.06) | 0.15 (0.20) | 0.07 (0.10) | 0.11 (0.14)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Alternative hypothesis was senofilcon A toric was superior to balafilcon A toric by having a lower logMAR score; Test type: Superiority or Other; p = 0.0083, t-test, 1 sided; Mean Difference (Final Values) = -0.13, Standard Deviation 0.15 — Mean difference was senofilcon A minus balafilcon A
Statistical Analysis 2: Comparison: Senofilcon A Toric vs Lotrafilcon B Toric; Alternative hypothesis was senofilcon A toric was superior to lotrafilcon B toric by having a lower logMAR score; Test type: Superiority or Other; p = 0.052, t-test, 1 sided; Mean Difference (Final Values) = -0.06, Standard Deviation 0.09 — Mean difference was senofilcon A minus lotrafilcon B
Statistical Analysis 3: Comparison: Senofilcon A Toric vs Omafilcon A Toric; Alternative hypothesis was senofilcon A toric was superior to omafilcon A toric by having a lower logMAR score; Test type: Superiority or Other; p = 0.015, t-test, 1 sided; Mean Difference (Final Values) = -0.13, Standard Deviation 0.14 — Mean difference was senofilcon A minus omafilcon A

3. Secondary Outcome: Degree of Lens Rotation in Superior Gaze.
Description: Degree of lens rotation while participant is gazing up.
Time Frame: After each of the four lens insertions
Population: Only participants who completed the study per protocol. Some participants had missing data for some lenses.
Measure: Mean (Standard Deviation); unit: Degree of rotation
Arm/Group | Senofilcon A Toric | Balafilcon A Toric | Lotrafilcon B Toric | Omafilcon A Toric
Number analyzed (Participants) | 13 | 13 | 13 | 11
Degree of rotation | 3.3 (3.8) | 6.0 (4.7) | 3.7 (2.6) | 6.5 (7.0)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Test type: Superiority or Other; p = 0.16, t-test, 1 sided; Mean Difference (Final Values) = -2.7, Standard Deviation 6.5 — Mean difference is senofilcon A minus balafilcon A
Statistical Analysis 2: Comparison: Senofilcon A Toric vs Lotrafilcon B Toric; Test type: Superiority or Other; p = 0.73, t-test, 1 sided; Mean Difference (Final Values) = -0.3, Standard Deviation 3.5 — Mean difference is senofilcon A minus lotrafilcon B
Statistical Analysis 3: Comparison: Senofilcon A Toric vs Omafilcon A Toric; Test type: Superiority or Other; p = 0.044, t-test, 1 sided; Mean Difference (Final Values) = -3.3, Standard Deviation 4.4 — Mean difference was senofilcon A minus omafilcon A

4. Secondary Outcome: Degree of Lens Rotation in Superior-temporal Gaze.
Description: Degree of lens rotation while participant is gazing up and out(towards the temple).
Time Frame: After each of 4 lens insertions.,
Population: Only participants who completed the study per protocol. Some participants had missing data for some lenses.
Measure: Mean (Standard Deviation); unit: Degree of rotation
Arm/Group | Senofilcon A Toric | Balafilcon A Toric | Lotrafilcon B Toric | Omafilcon A Toric
Number analyzed (Participants) | 13 | 13 | 13 | 11
Degree of rotation | 6.3 (5.5) | 9.4 (5.4) | 4.9 (2.3) | 8.6 (5.8)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Test type: Superiority or Other; p = 0.044, t-test, 1 sided; Median Difference (Final Values) = -3.1, Standard Deviation 5.0 — Mean difference is senofilcon A minus balafilcon A
Statistical Analysis 2: Comparison: Senofilcon A Toric vs Lotrafilcon B Toric; Test type: Superiority or Other; p = 0.31, t-test, 1 sided; Mean Difference (Final Values) = 1.4, Standard Deviation 4.7 — Mean difference is senofilcon A minus lotrafilcon B
Statistical Analysis 3: Comparison: Senofilcon A Toric vs Omafilcon A Toric; Test type: Superiority or Other; p = 0.44, t-test, 1 sided; Mean Difference (Final Values) = -1.5, Standard Deviation 5.9 — Mean difference is senofilcon A minus omafilcon A

5. Secondary Outcome: Degree of Lens Rotation in Superior-nasal Gaze.
Description: Degree of lens rotation while participant is gazing up and in(towards the nose).
Time Frame: After each of the four lens insertions
Population: Only participants who completed the study per protocol. Some participants had missing data for some lenses.
Measure: Mean (Standard Deviation); unit: Degree of rotation
Arm/Group | Senofilcon A Toric | Balafilcon A Toric | Lotrafilcon B Toric | Omafilcon A Toric
Number analyzed (Participants) | 13 | 13 | 13 | 11
Degree of rotation | 6.2 (5.4) | 5.6 (3.6) | 6.9 (4.8) | 5.8 (4.9)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Test type: Superiority or Other; p = 0.78, t-test, 1 sided; Mean Difference (Final Values) = 0.5, Standard Deviation 6.5 — Mean difference is senofilcon A minus balafilcon A
Statistical Analysis 2: Comparison: Senofilcon A Toric vs Lotrafilcon B Toric; Test type: Superiority or Other; p = 0.68, t-test, 1 sided; Mean Difference (Final Values) = -0.7, Standard Deviation 6.3 — Mean difference is senofilcon A minus lotrafilcon B
Statistical Analysis 3: Comparison: Senofilcon A Toric vs Omafilcon A Toric; Test type: Superiority or Other; p = 0.78, t-test, 1 sided; Mean Difference (Final Values) = -0.4, Standard Deviation 7.6 — Mean difference is senofilcon A minus omafilcon A

6. Secondary Outcome: Degree of Lens Rotation in Temporal Gaze.
Description: Degree of lens rotation while participant is gazing out(towards the temple).
Time Frame: After each of the four lens insertions
Population: Only participants who completed the study per protocol. Some participants had missing data for some lenses.
Measure: Mean (Standard Deviation); unit: Degree of rotation
Arm/Group | Senofilcon A Toric | Balafilcon A Toric | Lotrafilcon B Toric | Omafilcon A Toric
Number analyzed (Participants) | 13 | 13 | 13 | 11
Degree of rotation | 4.1 (3.1) | 7.2 (5.8) | 2.8 (2.2) | 6.6 (5.4)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Test type: Superiority or Other; p = 0.11, t-test, 1 sided; Mean Difference (Final Values) = -3.1, Standard Deviation 6.5 — Mean difference is senofilcon A minus balafilcon A
Statistical Analysis 2: Comparison: Senofilcon A Toric vs Lotrafilcon B Toric; Test type: Superiority or Other; p = 0.31, t-test, 1 sided; Mean Difference (Final Values) = 1.3, Standard Deviation 4.3 — Mean difference is senofilcon A minus lotrafilcon B
Statistical Analysis 3: Comparison: Senofilcon A Toric vs Omafilcon A Toric; Test type: Superiority or Other; p = 0.16, t-test, 1 sided; Median Difference (Final Values) = -3.0, Standard Deviation 6.3 — Mean difference is senofilcon A minus omafilcon A

7. Secondary Outcome: Degree of Lens Rotation in Nasal Gaze.
Description: Degree of lens rotation while participant is gazing in(towards the nose).
Time Frame: After each of the four lens insertions
Population: Only participants who completed the study per protocol. Some participants had missing data for some lenses.
Measure: Mean (Standard Deviation); unit: Degree of rotation
Arm/Group | Senofilcon A Toric | Balafilcon A Toric | Lotrafilcon B Toric | Omafilcon A Toric
Number analyzed (Participants) | 13 | 13 | 13 | 11
Degree of rotation | 3.2 (3.3) | 7.1 (5.9) | 2.4 (1.3) | 3.3 (3.2)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Test type: Superiority or Other; p = 0.061, t-test, 1 sided; Mean Difference (Final Values) = -3.9, Standard Deviation 6.8 — Mean difference is senofilcon A minus balafilcon A
Statistical Analysis 2: Comparison: Senofilcon A Toric vs Lotrafilcon B Toric; Test type: Superiority or Other; p = 0.47, t-test, 1 sided; Mean Difference (Final Values) = 0.8, Standard Deviation 3.9 — Mean difference is senofilcon A minus lotrafilcon B
Statistical Analysis 3: Comparison: Senofilcon A Toric vs Omafilcon A Toric; Test type: Superiority or Other; p = 0.38, t-test, 1 sided; Mean Difference (Final Values) = -1.0, Standard Deviation 3.6 — Mean difference is senofilcon A minus omafilcon A

8. Secondary Outcome: Degree of Lens Rotation Inferior-temporal Gaze.
Description: Degree of lens rotation while participant is gazing down and out.
Time Frame: After each of the four lens insertions
Population: Only participants who completed the study per protocol. Some participants had missing data for some of the lenses.
Measure: Mean (Standard Deviation); unit: Degree of rotation
Arm/Group | Senofilcon A Toric | Balafilcon A Toric | Lotrafilcon B Toric | Omafilcon A Toric
Number analyzed (Participants) | 13 | 13 | 13 | 11
Degree of rotation | 3.9 (3.9) | 5.3 (4.1) | 3.7 (2.8) | 2.5 (2.3)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Test type: Superiority or Other; p = 0.17, t-test, 1 sided; Mean Difference (Final Values) = -1.4, Standard Deviation 3.5 — Mean difference is senofilcon A minus balafilcon A
Statistical Analysis 2: Comparison: Senofilcon A Toric vs Lotrafilcon B Toric; Test type: Superiority or Other; p = 0.89, t-test, 1 sided; Mean Difference (Final Values) = 0.2, Standard Deviation 5.0 — Mean difference is senofilcon A minus lotrafilcon B
Statistical Analysis 3: Comparison: Senofilcon A Toric vs Omafilcon A Toric; Test type: Superiority or Other; p = 0.56, t-test, 1 sided; Mean Difference (Final Values) = 1.1, Standard Deviation 5.8 — Mean difference is senofilcon A minus omafilcon A

9. Secondary Outcome: Degree of Lens Rotation in Inferior-nasal Gaze.
Description: Degree of lens rotation while participant is gazing down and in.
Time Frame: After each of the four lens insertions
Population: Only participants who completed the study per protocol. Some participants had missing data for some of the lenses.
Measure: Mean (Standard Deviation); unit: Degree of rotation
Arm/Group | Senofilcon A Toric | Balafilcon A Toric | Lotrafilcon B Toric | Omafilcon A Toric
Number analyzed (Participants) | 13 | 13 | 13 | 11
Degree of rotation | 3.0 (1.6) | 9.0 (6.9) | 5.9 (2.9) | 9.5 (5.8)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Test type: Superiority or Other; p = 0.0080, t-test, 1 sided; Mean Difference (Final Values) = -6.0, Standard Deviation 6.8 — Mean difference is senofilcon A minus balafilcon A
Statistical Analysis 2: Comparison: Senofilcon A Toric vs Lotrafilcon B Toric; Test type: Superiority or Other; p = 0.0049, t-test, 1 sided; Mean Difference (Final Values) = -2.9, Standard Deviation 3.1 — Mean difference is senofilcon A minus lotrafilcon B
Statistical Analysis 3: Comparison: Senofilcon A Toric vs Omafilcon A Toric; Test type: Superiority or Other; p = 0.0058, t-test, 1 sided; Mean Difference (Final Values) = -6.4, Standard Deviation 5.6 — Mean difference is senofilcon A minus omafilcon A

10. Secondary Outcome: Degree of Lens Rotation in Inferior Gaze.
Description: Degree of lens rotation while participant is gazing down.
Time Frame: After each of the four lens insertions
Population: Only participants who completed the study per protocol. Some participants had missing data for some of the lenses.
Measure: Mean (Standard Deviation); unit: Degree of rotation
Arm/Group | Senofilcon A Toric | Balafilcon A Toric | Lotrafilcon B Toric | Omafilcon A Toric
Number analyzed (Participants) | 13 | 13 | 13 | 11
Degree of rotation | 3.9 (4.3) | 5.0 (4.0) | 4.2 (6.3) | 2.4 (1.9)
Statistical Analysis 1: Comparison: Senofilcon A Toric vs Balafilcon A Toric; Test type: Superiority or Other; p = 0.27, t-test, 1 sided; Mean Difference (Final Values) = -1.2, Standard Deviation 3.7 — Mean difference is senofilcon A minus balafilcon A
Statistical Analysis 2: Comparison: Senofilcon A Toric vs Lotrafilcon B Toric; Test type: Superiority or Other; p = 0.85, t-test, 1 sided; Mean Difference (Final Values) = -0.3, Standard Deviation 6.0 — Mean difference is senofilocon A minus lotrafilcon B
Statistical Analysis 3: Comparison: Senofilcon A Toric vs Omafilcon A Toric; Test type: Superiority or Other; p = 0.73, t-test, 1 sided; Mean Difference (Final Values) = 0.3, Standard Deviation 2.6 — Mean difference is senofilcon A minus omifilcon A

ADVERSE EVENTS:
Arm/Group | Lotrafilcon B / Senofilcon A / Balafilcon A / Omafilcon A | Lotrafilcon B / Omafilcon A / Senofilcon A / Balafilcon A | Lotrafilcon B / Balafilcon A / Senofilcon A / Omafilcon A | Senofilcon A / Lotrafilcon B / Omafilcon A / Balafilcon A | Senofilcon A / Omafilcon A / Balafilcon A / Lotrafilcon B | Senofilcon A / Balafilcon A / Lotrafilcon B / Omafilcon A | Omafilcon A / Lotrafilcon B / Senofilcon A / Balafilcon A | Balafilcon A / Lotrafilcon B / Senofilcon A / Omafilcon A | Balafilcon A / Lotrafilcon B / Omafilcon A / Senofilcon A | Balafilcon A / Senofilcon A / Lotrafilcon B / Omafilcon A | Balafilcon A / Senofilcon A / Omafilcon A / Lotrafilcon A | Balafilcon A / Omafilcon A / Lotrafilcon B / Senofilcon A
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.